CLINICAL TRIAL: NCT01105910
Title: Efficacy of Systane Ultra in Post Menopausal Women With Dry Eye
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: SMA-09-21
Record Dates: First submitted 2010-04-15; First posted 2010-04-19 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2012-01

CONDITIONS: Post Menopausal Dry Eye Subjects
Keywords: Dry Eye, Post Menopausal dry eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Systane Ultra (Experimental): Systane Ultra Lubricant Eye Drops
  Interventions: Other: Systane Ultra Lubricant Eye Drops
- Sensitive Eyes (Active Comparator): Sensitive Eyes Eye Drops (Bausch & Lomb)
  Interventions: Other: Sensitive Eyes Eye Drops (Bausch & Lomb)

INTERVENTIONS:
Other: Systane Ultra Lubricant Eye Drops — 1 to 2 drops in each eye 4 times per day for 30 days
  Arms: Systane Ultra
Other: Sensitive Eyes Eye Drops (Bausch & Lomb) — 1 to 2 drops in each eye 4 times per day for 30 days
  Arms: Sensitive Eyes

SUMMARY:
To evaluate the efficacy of Systane Ultra in post menopausal women with dry eye.

ELIGIBILITY:
Inclusion Criteria:

1. Post-menopausal (menses ceased more than 12 months prior to the start of the study).
2. Diagnosed for dry eye

Exclusion Criteria:

1. History of Sjögren's Syndrome or evidence of chronic dry eye syndrome. Confirmed autoimmune connective tissue diseases such as rheumatoid arthritis, fibromyalgia or scleroderma.
2. Active and severe blepharitis, rosacea and associated ocular sequelae.
3. Has any significant eyelid abnormality affecting lid function.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2010-02; Primary Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Reduction in corneal staining | 30 days

SECONDARY OUTCOMES:
Patient acceptability / comfort | 30 days

REFERENCES:
- [Result] http://www.aaopt.org/efficacy-evaluation-systane-ultra-lubricant-eye-drops-postmenopausal-women-dry-eye